CLINICAL TRIAL: NCT05986344
Title: Correlation Between Uterine Artery Doppler Indices and Menstrual Changes After Insertion of Copper Intrauterine Contraceptive Device and Levonorgestrel Intrauterine System
Brief Title: Uterine Artery Doppler and Menstrual Changes After Insertion Intrauterine Contraceptive Device
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, principle investigator/Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Other Study IDs: Doppler IUD
Record Dates: First submitted 2023-07-25; First posted 2023-08-14 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Intrauterine Contraceptive Device Complication
Keywords: Intrauterine Contraceptive Device; Doppler

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Copper intrauterine contraceptive device: Women will have the copper T-380 IUD (silverline, imported by DKT Egypt LLC-Egypt) ® IUD.
  Interventions: Device: Copper intrauterine contraceptive device
- Levonorgestrel Intrauterine System: Women will recieve the LNG-IUS (Mirena, Bayer HealthCare, Berlin, Germany)® IUD .
  Interventions: Device: LNG-IUS

INTERVENTIONS:
Device: Copper intrauterine contraceptive device — copper T-380 IUD
  Other Names: silverline
  Groups: Copper intrauterine contraceptive device
Device: LNG-IUS — Levonorgestrel Intrauterine System
  Other Names: mirena
  Groups: Levonorgestrel Intrauterine System

SUMMARY:
To evaluate the correlation between uterine artery Doppler indices and subsequent menstrual changes after 3 months of insertion of copper T-380 IUD and LNG-IUS

DETAILED DESCRIPTION:
A randomized prospective clinical trial

Study Population:

The study population includes multiparous women, having normal menstrual cycles, who are eligible for insertion of IUCD. Women will be recruited for enrollment when they come to the family planning clinic. They will be counseled about different contraceptive options. If they want to have the IUCD, they will be asked to participate in the study after been evaluated to ensure fulfilling inclusion and exclusion criteria Women will be enrolled in the study after giving written informed consent Group (A): ….Women will have the copper T-380 IUD (PREGNA, India, imported by DKT Egypt LLC-Egypt) ® IUD.

Group (B): …. Women will recieve the LNG-IUS (Mirena, Bayer HealthCare, Berlin, Germany)® IUD .

ELIGIBILITY:
Inclusion Criteria:

* Desire to have intrauterine contraceptive device after counseling about different contraceptive options and consented to the study.
* Normal menstrual bleeding cycles (24-35 days).

Exclusion Criteria:

1. Nulliparity.
2. Undiagnosed uterine bleeding.
3. Any proven ovarian, uterine or endometrial pathology such as; uterine myoma, adenomyosis, endometrial polyps, ovarian cysts
4. Contraceptive pills had not been taken during the previous 3 months and any previous IUD had been removed at least 1 month earlier
5. Hemorrhagic disorders.
6. Acute or chronic pelvic inflammatory disease
7. Known uterine anomalies e.g., Bicornuate/septate Uterus.
8. Anemia (hemoglobin <10 g/dl).
9. Diagnosis of active cervical infection
10. Dysplasia in the cervix.
11. Patients wishing post-partum or post-abortum IUD insertion

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population includes multiparous women, having normal menstrual cycles, who are eligible for insertion of IUCD. Women will be recruited for enrollment when they come to the family planning clinic. They will be counseled about different contraceptive options. If they want to have the IUCD, they will be asked to participate in the study after been evaluated to ensure fulfilling inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
menstrual changes. | 3 months after insertion
  Pictorial blood loss assessment chart PBAC score (a score >100was equivalent to blood loss >80 mL)
uterine artery pulsatility index | 3 months after insertion
  trans-vaginal ultrasound pulsed doppler

CONTACTS AND LOCATIONS:
Overall Officials: Beni-Suef University, Principal Investigator — Faculty of Medicine Beni-Suef University
Locations (1):
- Beni-suef university Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided